CLINICAL TRIAL: NCT04260841
Title: Passive Leg Raising 3.0 and Fluid Responsiveness
Brief Title: Passive Leg Raising and Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, research coordinator, Frisius Medisch Centrum
Other Study IDs: nWMO 217
Record Dates: First submitted 2017-06-09; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Passive Leg Raising
Keywords: fluid responsiveness
MeSH Terms: interventions — Beds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: bed in 45 degrees for passive leg raising test — fluid responsiveness is tested by the passive leg raising test
  Other Names: use of "pillow" for passive leg raising test

SUMMARY:
In the Intensive Care the Passive Leg Raising (PLR) test is a validated instrument to predict fluid responsiveness. In this study the investigators will try to prove the similarity of PLR test with a pillow and the PLR test with the patients bed in 45 degrees.

DETAILED DESCRIPTION:
PLR test with pillow PLR test with bed to avoid a difference in results by the order of the measurements, the order of PLR testing is random.

ELIGIBILITY:
Inclusion Criteria:

* admission on Intensive Care
* clinical signs as; mean arterial pressure < 60, lactate > 2.0 mmol/L

Exclusion Criteria:

* age < 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with clinical signs of fluid need
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
fluid responsiveness expressed in volume | from ICU admission until ICU discharge; test performed on the moment of clinical signs of fluid need through study completion, an average of 5 days
  are both PLR tests similar / comparable on fluid responsiveness
blood pressure expressed in mmHg | test performed on the moment of clinical signs of fluid need through study completion, an average of 5 days
  are both PLR tests similar / comparable on fluid responsiveness
cardiac output | test performed on the moment of clinical signs of fluid need through study completion, an average of 5 days
  are both PLR tests similar / comparable on fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — MCL
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No